CLINICAL TRIAL: NCT07340541
Title: TBCRC Evolutionary Clinical Trial for Novel Biomarker-Driven Therapies (EVOLVE-BDT)
Brief Title: Evolutionary Clinical Trial for Novel Biomarker-Driven Therapies
Acronym: EVOLVE-BDT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: Advanced Research Projects Agency for Health (ARPA-H) (Unknown); Breast Cancer Research Foundation (Other); Translational Breast Cancer Research Consortium (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LCCC2521-PARENT/TBCRC-073; 140D042590009 (Other: ARPA-H)
Record Dates: First submitted 2026-01-12; First posted 2026-01-14 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; Triple Negative Breast Cancer; Estrogen-receptor-positive Breast Cancer; Hormone Receptor Negative Breast Carcinoma
Keywords: biomarker directed therapies; biomarker stratified trial
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — abemaciclib; Everolimus; Capecitabine; Androgen Antagonists

STUDY DESIGN:
Intervention Model Description: Patients are stratified according to tumor marker profiles and receive corresponding treatment regimens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Cohort 1 Arm A (Experimental): ER+ (Estrogen Receptor Positive) and HER2- (Human Epidermal Growth Factor Receptor 2 Negative). ESR1 mutant positive or negative and Phosphatidylinositol 3-kinase catalytic subunit alpha / AKT serine/threonine kinase / PTEN loss or deletion negative.
  Interventions: Drug: SERD* + abemaciclib
- Cohort 1- Arm B (Experimental): ER+ (Estrogen Receptor Positive) and HER2- (Human Epidermal Growth Factor Receptor 2 Negative). ESR1 mutant positive or negative and Phosphatidylinositol 3-kinase catalytic subunit alpha / AKT serine/threonine kinase / PTEN loss or deletion negative.
  Interventions: Drug: SERD* + everolimus
- Cohort 2 Arm A (Experimental): ER+ (Estrogen Receptor Positive) and HER2- (Human Epidermal Growth Factor Receptor 2 Negative). ESR1 mutant negative or positive, and Phosphatidylinositol 3-kinase catalytic subunit alpha / AKT serine/threonine kinase / PTEN loss or deletion positive.
  Interventions: Drug: SERD* + abemaciclib
- Cohort 2 Arm B (Experimental): ER+ (Estrogen Receptor Positive) and HER2- (Human Epidermal Growth Factor Receptor 2 Negative). ESR1 mutant negative or positive, and Phosphatidylinositol 3-kinase catalytic subunit alpha / AKT serine/threonine kinase / PTEN loss or deletion positive.
  Interventions: Drug: SERD* + everolimus or capecitabine
- Cohort 3 (Active Comparator): Triple-Negative Breast Cancer (TNBC): ER- (Estrogen receptor negative), PR- (Progesterone receptor negative), HER2- HER2 negative. AR - = Androgen Receptor negative, PD-L1 (Programmed Death-Ligand 1) positive or negative.
  Interventions: Drug: SOC
- Cohort 4 (Experimental): Triple-Negative Breast Cancer (TNBC): ER- (Estrogen receptor negative), PR- (Progesterone receptor negative), HER2- HER2 negative. AR + = Androgen Receptor positive, PD-L1 (Programmed Death-Ligand 1) positive or negative.
  Interventions: Drug: Antiandrogen

INTERVENTIONS:
Drug: SERD* + abemaciclib — Investigators choice Selective Estrogen Receptor Degrader + abemaciclib therapy.
  Arms: Cohort 1 Arm A; Cohort 2 Arm A
Drug: SERD* + everolimus — Investigators choice Selective Estrogen Receptor Degrader + everolimus therapy.
  Arms: Cohort 1- Arm B
Drug: SERD* + everolimus or capecitabine — Investigators choice Selective Estrogen Receptor Degrader + everolimus or capecitabine therapy.
  Arms: Cohort 2 Arm B
Drug: SOC — standard-of-care (SOC) chemotherapy in breast cancer
  Arms: Cohort 3
Drug: Antiandrogen — Antiandrogen therapy
  Arms: Cohort 4

SUMMARY:
This is a multicenter, multi-arm, biomarker-stratified trial designed to evaluate biomarker-directed therapies in patients with estrogen receptor-positive/hormone receptor-negative (ER+/HR-) and triple-negative (TN) metastatic breast cancer (MBC). The trial integrates both retrospective and prospective data collection, including archival tumor tissue, medical record abstraction, and prospective tumor and blood sampling prior to initiation of protocol directed treatment. Based on biomarker subtype, participants will receive standard of care therapy. Liquid biopsy will be collected on Cycle 2 Day 1, and then liquid biopsy, imaging and clinical data will be collected at each re-staging. Treatment will continue until discontinuation for progression, toxicity or at the discretion of the treating physician.

DETAILED DESCRIPTION:
The platform design makes it easy to assess multiple targeted therapies at the same time, focusing on patient groups identified by specific biomarkers. Patients who experience disease progression may be reassigned to additional eligible sub trials evaluating alternative therapeutic options. The primary endpoint for each arm is progression-free survival (PFS). This adaptive framework enables continuous learning and rapid translation of biomarker discoveries into therapeutic evaluation, promoting an agile and data-driven approach to treatment optimization in advanced breast cancer.

Beyond ER and HER2, there are few biomarkers to drive treatment decisions in metastatic and primary breast cancer, leaving a gap in effective treatments for other subtypes. To address this, triple-negative (TNBC) is pioneering an adaptive, evolutionary trial focusing on women with metastatic breast cancer (MBC) in the second-line (2L) setting. The adaptive trial infrastructure is designed to serve as an integrated parent study, enabling coordinated acquisition of clinical and translational data, as well as training and testing activities. Within this framework, individual biomarker-driven sub-trials (based on biomarker development) can be created and conducted.

Eligible participants include patients with ER+/HER2- or triple-negative (TNBC) metastatic breast cancer (MBC) who have progressed on first line (1L) therapy but have not yet initiated second-line (2L) treatment. HER2+ patients will be excluded due to the availability of established effective therapies.

This Sub Protocol #1 will enroll subjects based on biomarker subtype. Participants will receive a standard of care therapy. Liquid biopsy will be collected on Cycle 2 Day 1, and then liquid biopsy, imaging and clinical data will be collected at each re-staging. Treatment will continue until discontinuation for progression, toxicity or at the discretion of the treating physician. In order to participate in Sub Protocol #1 subjects must have consented to the Parent protocol.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained to participate in the study and HIPAA authorization for release of personal health information.
* Subject is willing and able to comply with study procedures based on the judgement of the investigator.
* Age ≥ 18 years of age at the time of consent
* ECOG Performance Status of 0-2 (see APPENDIX A: ECOG Performance Status Scale).
* Patients must fulfill all eligibility criteria outlined in the LCCC2521 Parent Protocol and consented to LCCC2521 Parent Protocol

Exclusion Criteria:

* Inaccessible metastatic lesion to research biopsy
* Subject has already initiated 2nd line therapy
* Concurrent disease or condition that in the opinion of the treating oncologist renders the patient inappropriate for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-06-02 (Estimated); Study Completion 2028-06-02 (Estimated)

PRIMARY OUTCOMES:
Intra-Individual Progression-Free Survival (PFS) | Up to 5 years
  Progression-Free Survival (PFS) is defined as the time from initiation of study therapy until documented disease progression per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1 or death from any cause, whichever occurs first. For intra-individual comparisons across successive therapy lines, a PFS ratio will be calculated by dividing the PFS of the current line (nth line, PFSₙ) by the PFS of the preceding line ((n-1)th line, PFSn-1). This allows each patient to serve as their own control, reducing between-patient variability and normalizing for the expected decline in PFS with later lines. RECIST v1.1 defines Complete Response (CR) as disappearance of all target lesions, Partial Response (PR) as ≥30% decrease, Stable Disease (SD) as insufficient change for PR or PD, and Progressive Disease (PD) as ≥20% increase, measurable growth in non-target lesions, or new lesions.
Progression free survival (PFS) -Within Arm Evaluation | Up to 5 years
  This endpoint assesses PFS in a specific treatment arm compared with a prespecified historical control derived from contemporary real-world data or prior clinical trials. Progression-Free Survival (PFS) is defined as the time from initiation of study therapy until documented disease progression per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1 or death from any cause, whichever occurs first. RECIST v1.1 defines Complete Response (CR) as disappearance of all target lesions, Partial Response (PR) as ≥30% decrease, Stable Disease (SD) as insufficient change for PR or PD, and Progressive Disease (PD) as ≥20% increase, measurable growth in non-target lesions, or new lesions.

SECONDARY OUTCOMES:
Progression free survival (PFS) - Between-Arm Evaluation | Up to 3 months
  This endpoint assesses between two or more concurrently accruing arms, typically an investigational or biomarker-driven regimen versus a shared control or reference arm. Progression-Free Survival (PFS) is defined as the time from initiation of study therapy until documented disease progression per Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1 or death from any cause, whichever occurs first. RECIST v1.1 defines Complete Response (CR) as disappearance of all target lesions, Partial Response (PR) as ≥30% decrease, Stable Disease (SD) as insufficient change for PR or PD, and Progressive Disease (PD) as ≥20% increase, measurable growth in non-target lesions, or new lesions.
Tissue- and blood-based biomarkers on response rate | Up to 3 months
  Tissue- and blood-based biomarkers predictive of response or resistance to standard-of-care first- and second-line therapies will be investigated. Response Evaluation Criteria In Solid Tumors Criteria (RECIST) v1.1 will be used for tumor response assessment. RECIST v1.1 defines Complete Response (CR) as disappearance of all target lesions, Partial Response (PR) as ≥30% decrease, Stable Disease (SD) as insufficient change for PR or PD, and Progressive Disease (PD) as ≥20% increase, measurable growth in non-target lesions, or new lesions.
Overall survival (OS) | Up to 12 months
  Overall survival (OS) is defined as the time from initiation of study therapy to death from any cause.
Objective response rate (ORR) | Up to 3 months
  Objective response rate (ORR) is defined as the proportion of subjects with a complete response or partial response to treatment according to Response Evaluation Criteria in Solid Tumors (RECIST)v1.1. RECIST v1.1 defines Complete Response (CR) as disappearance of all target lesions, Partial Response (PR) as ≥30% decrease, Stable Disease (SD) as insufficient change for PR or PD, and Progressive Disease (PD) as ≥20% increase, measurable growth in non-target lesions, or new lesions.
Duration of response (DoR) | Up to 12 months
  DOR is defined as the time from documentation of PR or better to progressive disease (PD) and will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 for each investigational regimen. RECIST v1.1 defines Complete Response (CR) as disappearance of all target lesions, Partial Response (PR) as ≥30% decrease, Stable Disease (SD) as insufficient change for PR or PD, and Progressive Disease (PD) as ≥20% increase, measurable growth in non-target lesions, or new lesions.
Clinical benefit rate (CBR) | Up to 12 months
  Clinical benefit rate (CBR) is defined as the proportion of patients who achieve a complete response (CR), partial response (PR), or stable disease (SD) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. RECIST v1.1 defines Complete Response (CR) as disappearance of all target lesions, Partial Response (PR) as ≥30% decrease, Stable Disease (SD) as insufficient change for PR or PD, and Progressive Disease (PD) as ≥20% increase, measurable growth in non-target lesions, or new lesions. C
Grade 2 or above Adverse Events per NCI Common Terminology Criteria for Adverse Events (CTCAE) | Up to 12 months
  Grade 2 or above treatment attributed Adverse Events per NCI CTCAE will be reported. The NCI CTCAE is a descriptive terminology which can be utilized for Adverse Event (AE) reporting. A grading (severity) scale is provided for each AE term. Grade 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated. Grade 2 Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental Activities of Daily Living (ADL). Grade 3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Grade 4 Life-threatening consequences; urgent intervention indicated. Grade 5 Death related to AE.
Changes in circulating tumor DNA (ctDNA) levels | Up to 12 months
  Changes in circulating tumor DNA (ctDNA) levels and mutation profiles under therapeutic pressure over time will be assessed. Circulating tumor DNA (ctDNA) mutation profiles during treatment will be assessed via blood draws using the Tempus Xf assay. Detected set of oncogenic drivers, resistance mutations, single nucleotide variants (SNVs), insertions and deletions (INDELs), copy number gains (CNGs) and gene rearrangements will be reported.
Changes in transcriptomic data - tissue | Up to 12 months
  Changes in transcriptomic profiles under therapeutic pressure will be assessed over time. Transcriptomic data from baseline and post-baseline primary or metastatic tumor tissue will be generated using the Tempus XR platform, providing quantitative gene expression levels for each panel gene per sample.
Changes in transcriptomic data - blood | Up to 12 months
  Transcriptomic changes under therapeutic pressure will be assessed over time using evRNA-seq expression levels obtained from blood-derived extracellular vesicles, in patient blood will provide quantitative estimates of gene transcript levels transcriptome-wide.
Changes in Circulating tumor DNA (ctDNA) and tumor response relation | Up to 12 months
  Changes in ctDNA and tumor response relation over time will be assessed. ctDNA will be assessed via blood draws using the Tempus Xf assay and gene rearrangements will be reported. Tumor response will be evaluated at corresponding time points using RECIST v1.1 criteria. RECIST v1.1 defines Complete Response (CR) as disappearance of all target lesions, Partial Response (PR) as ≥30% decrease, Stable Disease (SD) as insufficient change for PR or PD, and Progressive Disease (PD) as ≥20% increase, measurable growth in non-target lesions, or new lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A Carey, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center; Eric Winer, MD, Study Chair — Yale University
Locations (1):
- Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials